CLINICAL TRIAL: NCT03161158
Title: PURE-HF: Peripheral Ultrafiltration for the RElief From Congestion in Heart Failure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Fresenius Medical Care Deutschland GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF-HF-02-INT; EUDAMED-No. CIV -17-01-018204 (Other: European Medicines Agency)
Record Dates: First submitted 2017-05-02; First posted 2017-05-19 (Actual); Results first posted 2021-05-05 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2020-07

CONDITIONS: Heart Failure; Acute Heart Failure
Keywords: Cardio-Renal Syndrome type 1; Acutely decompensated chronic heart failure; Ultrafiltration
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, randomized, parallel-group, controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrafiltration Group (Active Comparator): Veno-venous ultrafiltration (CHIARA-System) complementary to low-dose diuretic therapy according to treatment algorithm.
  Interventions: Device: CHIARA-System
- Control group (Usual care IV diuretics) (Other): Guideline-directed therapy including IV loop diuretics according to treatment algorithm.
  Interventions: Other: Usual care IV diuretics

INTERVENTIONS:
Device: CHIARA-System — Treatment with veno-venous ultrafiltration (CHIARA-System) complementary to low-dose diuretic therapy according to treatment algorithm. 1-7 Ultrafiltration sessions (6-10h/session, number of sessions depending on clinical assessment) for at least 1-2 consecutive days and a maximum of 7 days.
  Other Names: Low-dose IV diuretics
  Arms: Ultrafiltration Group
Other: Usual care IV diuretics — Guideline-directed therapy including IV loop diuretics (according to treatment algorithm)
  Arms: Control group (Usual care IV diuretics)

SUMMARY:
This study evaluates whether tailored, peripheral ultrafiltration complementary to low-dose diuretics is associated with a reduction in cardiovascular mortality in 90 days after randomization and heart failure events in 90 days after discharge than usual care including stepped intravenous diuretics in acutely decompensated chronic heart failure with fluid overload (not fully responsive to diuretic therapy).

DETAILED DESCRIPTION:
The study will evaluate whether stepped, peripheral ultrafiltration complementary to low-dose diuretics influences 90-day clinical outcomes compared to usual care including intravenous diuretics in symptomatic heart failure patients with persistent congestion. Hospitalized subjects will be randomly assigned to receive either a tailored, peripheral ultrafiltration approach complementary to intravenous low-dose diuretics and other guideline-directed medical therapy OR high-dose diuretic therapy and other Guideline-directed medical therapy.

ELIGIBILITY:
Inclusion Criteria:

General:

Informed consent signed and dated by study patient and investigator/authorised physician

* Minimum age of 18 years
* Ability to understand the nature and requirements of the study

Study-specific:

* Heart failure patients with preserved, mid-range or reduced ejection fraction (confirmed according to the current definitions of heart failure with preserved (HFpEF), mid-range (HFmrEF) and reduced ejection fraction (HFrEF) requiring echocardiographic assessment within the prior 12 months) who are admitted to the hospital due to signs/symptoms of congestion (left- or right sided)
* On regularly scheduled oral loop diuretics prior to admission
* Patients who have received IV loop diuretics for decongestion within 24 hours after hospital admission and prior to screening. The dosages are administered according to clinical judgment.** (**This inclusion criterion was changed with CIP amendment; in former version 3.0 it read "After pre-screening and prior to final screening for eligibility, patients who have received two boluses of IV loop diuretics (Dose according to the Furosemide-Low Intensification, Q12 hour bolus arm of the DOSE trial))
* Symptoms of congestion and clinical evidence at the time of final screening for eligibility:
* Fluid overload manifested by at least 2 of the following:

  1. Pitting edema ≥2+ of the lower extremities
  2. Jugular venous pressure >8 cm H2O
  3. Pulmonary congestion or pleural effusion on chest x-ray
  4. Paroxysmal nocturnal dyspnea or ≥2- pillow orthopnea
  5. Respiration rate ≥20 per minute
* Additional objective documentation of congestion: Lung or inferior vena cava ultrasound, chest x-ray or elevated filling pressures, if available, at the time of randomization (optional)

Exclusion Criteria:

General:

* Any condition which could interfere with the patient's ability to comply with the study
* In case of female patients, pregnancy or lactation period
* Participation in an interventional clinical study during the preceding 30 days
* Previous participation in the same study
* Unwillingness or inability to complete follow up
* Active drug or alcohol abuse (smoking allowed)

Study-specific:

* Acute coronary syndrome requiring intervention during index hospitalization
* Severe renal dysfunction requiring renal replacement therapy
* Systolic blood pressure < 90 mmHg at the time of randomization
* Pulmonary hypertension not secondary to left heart disease
* Pulmonary disease thought to be primarily responsible for symptoms
* Contraindication to systemic anticoagulation
* Severe concomitant disease expected to prolong hospitalization or to cause death in ≤ 90 days
* Sepsis
* Severe uncorrected valvular stenosis at the time of randomization
* Active myocarditis
* Hypertrophic obstructive cardiomyopathy
* Constrictive pericarditis or restrictive cardiomyopathy
* Liver cirrhosis due to primary liver disease* (*Restriction "due to primary liver disease" was present after amendment in study protocol version 5.0 but not in version 3.0)
* Known infection with human immunodeficiency virus (HIV) or active hepatitis C
* Previous solid organ transplant
* Presence or requirement for mechanical respiratory support
* Presence or requirement of a mechanical circulatory support device
* Need for IV positive inotropic agents at the time of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-11-03 (Actual); Primary Completion 2019-08-26 (Actual); Study Completion 2019-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Ruschitzka, Prof Dr med, Study Chair — Universitätsspital Zürich, Klinik für Kardiologie
Locations (11):
- Germany (6):
  - Universitätsklinikum Aachen (Med. Klinik II), Aachen
  - Helios Klinikum Duisburg, Duisburg
  - Helios Klinikum Erfurt GmbH, Erfurt
  - Medizinische Universitätsklinik, Innere Medizin III, Heidelberg
  - Helios Klinikum Hildesheim GmbH, Hildesheim
  - Klinikum Stuttgart, Klinik für Nieren-, Hochdruck- und Autoimmunerkrankungen, Stuttgart
- Sweden (5):
  - Falun Hospital, Falun
  - Universitetssjukhuset Örebro, Hjärtsviktsmottagningen, Örebro
  - Danderyds University Hospital, Stockholm
  - Karolinska University Hospital Huddinge, Department of Cardiology, Stockholm
  - Uppsala University Hospital, Department of Cardiology, Uppsala

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srivastava M, Harrison N, Caetano AFS, Tan AR, Law M. Ultrafiltration for acute heart failure. Cochrane Database Syst Rev. 2022 Jan 21;1(1):CD013593. doi: 10.1002/14651858.CD013593.pub2. PMID 35061249

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 62 enrolled patients, 44 were randomized to treatment. 37 patients were included in the safety and full analysis set (SAF/FAS)
Period: Overall Study
Arm/Group | Ultrafiltration Group | Control Group (Usual Care IV Diuretics)
Started (Patients in the FAS) | 18 | 19
Completed (Patients in the FAS) | 9 | 13
Not Completed | 9 | 6

BASELINE CHARACTERISTICS:
Population: Of 44 randomized patients, 37 were included in the safety and full analysis set (SAS/ FAS).
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrafiltration Group | Control Group (Usual Care IV Diuretics) | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (9.45) | 74.2 (12.40) | 72.9 (11)
Age, Customized [Count of Participants; unit: Participants]
  <45 years | 0 | 1 | 1
  ≥ 45 to <65 years | 6 | 2 | 8
  ≥65 years | 12 | 16 | 28
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 8
  Male | 15 | 14 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 18 | 19 | 37
Height [Mean (Standard Deviation); unit: cm] | 173.4 (7.80) | 172.3 (13.28) | 172.8 (10.83)
Weight [Mean (Standard Deviation); unit: kg] | 106.4 (33.17) | 95.6 (27.42) | 100.9 (30.42)
Body-Mass-Index (BMI) [Count of Participants; unit: Participants]
  ≥18.5 to <25 kg/m^2 | 1 | 4 | 5
  ≥25 to <30 kg/m^2 | 8 | 4 | 12
  ≥30 to <35 | 1 | 6 | 7
  ≥35 to <40 kg/m^2 | 2 | 3 | 5
  ≥40 kg/m^2 | 6 | 2 | 8
Systolic Blood Pressure (SBP) [Mean (Standard Deviation); unit: mmHg] | 117.6 (26.23) | 128.5 (29.84) | 123.2 (28.30)
Diastolic Blood Pressure (DBP) [Mean (Standard Deviation); unit: mmHg] | 68.4 (10.62) | 70.4 (14.68) | 69.4 (12.73)
Heart rate [Mean (Standard Deviation); unit: bpm] | 73.2 (20.32) | 71.9 (14.57) | 72.5 (17.28)
New York Heart Association (NYHA) Functional Classification [Count of Participants; unit: Participants] — The NYHA system classifies Heart Failure (HF) patients into four categories according to their symptons. Patients graded in NYHA class I show no limitation of physical activity, whereas patients graded in NYHA class IV are unable to carry on physical activity without discomfort.
  Participants
    NYHA I | 0 | 0 | 0
    NYHA II | 1 | 0 | 1
    NYHA III | 14 | 14 | 28
    NYHA IV | 2 | 5 | 7
    Missing | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Heart Failure (HF) Event
Description: Heart failure hospitalization or unscheduled outpatient or emergency department treatment with IV loop diuretics or ultrafiltration.
Time Frame: in 90 days after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrafiltration Group | Control Group (Usual Care IV Diuretics)
Number analyzed (Participants) | 18 | 19
Participants | 4 | 4

2. Primary Outcome: Cardiovascular Death up to 90 Days After Randomization.
Description: The rationale for the follow up time period of 90 days is that death rates reported in previous acute HF trials indicate that mortality seems to become linear after ~60-90 days post discharge Collection for Cardiovascular Trials initiative definition of cardiovascular death includes death resulting from an acute myocardial infarction, sudden cardiac death, death due to heart failure, death due to stroke, and death due to other cardiovascular causes
Time Frame: in 90 days after discharge
Measure: Count of Participants; unit: Participants
Arm/Group | Ultrafiltration Group | Control Group (Usual Care IV Diuretics)
Number analyzed (Participants) | 18 | 19
Participants | 4 | 1

ADVERSE EVENTS:
Time Frame: Per patient adverse events were collected from signed informed consent until max 30 days after last clinical Investigation visit.
Description: Adverse Event Definition and Collection has been according to ISO 14 155 "Clinical investigation of medical devices for human subjects - Good clinical practice."
Arm/Group | Ultrafiltration Group | Control Group (Usual Care IV Diuretics)
All-Cause Mortality (participants affected / at risk) | 7/18 | 2/19
Serious Adverse Events (participants affected / at risk) | 15/18 | 13/19
Other Adverse Events (participants affected / at risk) | 12/18 | 14/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrafiltration Group (N=18) | Control Group (Usual Care IV Diuretics) (N=19)
Cardiac Failure (Cardiac disorders) | 6 (6) | 4 (7)
Atrioventricular (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Cardiovascular (Cardiac disorders) | 1 (1) | 0 (0)
Sinoatrial block (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular (Cardiac disorders) | 0 (0) | 1 (1)
Acute kidney (Renal and urinary disorders) | 2 (2) | 2 (2)
Renal failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Nephrotic (Renal and urinary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Dementia (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Catheter (Surgical and medical procedures) | 1 (1) | 0 (0)
Stent placement (Surgical and medical procedures) | 0 (0) | 1 (1)
Abdominal wall (Gastrointestinal disorders) | 1 (1) | 0 (0)
Echocardiogram (Investigations) | 1 (1) | 0 (0)
Oxygen saturation (Investigations) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Device dislocation (Product Issues) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Loss of personal (Social circumstances) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ultrafiltration Group (N=18) | Control Group (Usual Care IV Diuretics) (N=19)
Oedema peripheral (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 2
Cyst (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Therapeutic product ineffective (General disorders) | 1 | 0
Vessel puncture site haematoma (General disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 3
Chronic kidney disease (Renal and urinary disorders) | 1 | 1
Haematuria (Renal and urinary disorders) | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1
Hypotension (Vascular disorders) | 3 | 2
Haematoma (Vascular disorders) | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 0
Wound (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 1
Escherichia infection (Infections and infestations) | 0 | 1
Escherichia urinary tract infection (Infections and infestations) | 0 | 1
Arthralgia (Metabolism and nutrition disorders) | 1 | 1
Back pain (Metabolism and nutrition disorders) | 2 | 0
Flank pain (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal pain (Metabolism and nutrition disorders) | 1 | 0
Pain in extremity (Metabolism and nutrition disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 1
Dementia Alzheimer's type (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Cardiac resynchronisation therapy (Surgical and medical procedures) | 1 | 0
Cardioversion (Surgical and medical procedures) | 1 | 0
Dialysis device insertion (Surgical and medical procedures) | 1 | 0
Percutaneous coronary intervention (Surgical and medical procedures) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 1 | 1
Decubitis ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Needle issue (Product Issues) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Due to the premature termination of the study and a resulting sample size of 37 patients in both analyses sets no statistical testing for any study endpoint has been applied. All study objectives were analyzed purely descriptively, continuous data with sample statistics, categorical data by frequency tables.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-19): https://cdn.clinicaltrials.gov/large-docs/58/NCT03161158/Prot_SAP_000.pdf